CLINICAL TRIAL: NCT04149860
Title: Interventional, Randomized, Double-blind, Placebo-controlled, Single-ascending-dose Study Investigating the Safety, Tolerability, and Pharmacokinetic Properties of Lu AF87908 in Healthy Subjects and Patients With Alzheimer's Disease
Brief Title: Study With Lu AF87908 in Healthy Participants and Participants With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 18146A
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Healthy; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Lu AF87908 or Placebo (Experimental): Participants in Cohorts A1 to A6 will receive a single dose of either Lu AF87908 or matching placebo at specific dose levels on Day 1.
  Interventions: Drug: Lu AF87908; Drug: Placebo
- Part B: Lu AF87908 or Placebo (Experimental): Participants in Cohorts B1 to B3 will receive a single dose of either Lu AF87908 or matching placebo at specific dose levels on Day 1.
  Interventions: Drug: Lu AF87908; Drug: Placebo
- Part C: Lu AF87908 or Placebo (Experimental): Participants in Cohorts C1 and C4 will receive a single dose of either Lu AF87908 or matching placebo at specific dose levels on Day 1.
  Interventions: Drug: Lu AF87908; Drug: Placebo

INTERVENTIONS:
Drug: Lu AF87908 — Lu AF87908 concentrate for solution for intravenous (IV) infusion
Drug: Placebo — Concentrate for solution for IV infusion

SUMMARY:
The purpose of this study is to investigate the safety of a single dose of Lu AF87908, how well it is tolerated and what the body does to the drug in healthy participants and participants with Alzheimer's disease.

DETAILED DESCRIPTION:
The study will be divided into three parts: Part A, Part B and Part C.

Part A consists of up to 6 sequential cohorts (Cohorts A1 to A6):

-Cohorts A1 to A6: 8 healthy participants per cohort (aiming for an equal number of men and women): 6 randomized to Lu AF87908 and 2 randomized to placebo.

Part B consists of up to 3 sequential cohorts (Cohorts B1 to B3):

-Cohorts B1 to B3: 4 Japanese and 4 Chinese healthy participants per cohort: 6 participants randomized to Lu AF87908 and 2 participants randomized to placebo.

Part C consists of 2 sequential cohorts (Cohorts C1 and C4):

-Cohort C1 will consist of 6 participants with Alzheimer's disease with 3:1 randomization scheme for active: placebo. Cohort C4 will consist of up to 8 participants. Cohort C4 participants will be randomized based on the randomization scheme from Cohort C1.

ELIGIBILITY:
Inclusion criteria

Healthy Participants:

-Men and women ≥18 and ≤65 years of age with a body mass index (BMI) ≥18 and ≤32 kilograms (kg)/square meter (m^2) and a minimum weight of 50 kg.

Participants with Alzheimer's disease:

* Men and women with a clinical diagnosis of Alzheimer's disease, Stages 3-4 according to the FDA guidelines.
* Mini-Mental State Examination (MMSE) of 15-30.
* Clinical Dementia Scale (CDR) global score up to and including 2.0.
* Confirmed or determined (via amyloid positron emission tomography [PET] scan) to be amyloid positive.
* If on FDA approved Alzheimer's disease medication, the treatment has been stable for 4 months prior to Day 1.

  -≥50 years of age.
* BMI ≥18 and ≤40 kg/m^2 and a minimum weight of 50 kg.

Exclusion criteria:

* Clinically relevant structural brain abnormality as assessed using magnetic resonance imaging (MRI).
* Any past or current treatment with an anti-Abeta or anti-tau active vaccine.
* Any past or current treatment with a monoclonal anti-tau antibody or a tau anti-sense oligomer within the last 6 months.
* Treatment with covid-19, influenza or pneumonia vaccine within the last 30 days prior to dosing of investigational medicinal product (IMP).

Other eligibility criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events | From Day 0 to Day 84
  Safety and tolerability based on the safety assessments (clinical safety laboratory tests, vital signs, weight, ECG parameters and physical examination)
AUC(0-t) of Lu AF87908 | From Day 0 to Day 84
  Area under the plasma concentration curve for Lu AF87908
Cmax of Lu AF87908 | From Day 0 to Day 84
  Maximum observed plasma concentration for Lu AF87908
Tmax Lu AF87908 | From Day 0 to Day 84
  Nominal time of occurrence of Cmax of Lu AF97908 in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (6):
- United States (6):
  - PAREXEL International, Glendale, California
  - Research Center of America, Hollywood, Florida
  - Panax Clinical Research, Miami, Florida
  - iResearch Atlanta LLC, Decatur, Georgia
  - Princeton Medical Institute, Princeton, New Jersey
  - Clinilabs, Inc., New York, New York

IPD SHARING:
Plan to Share IPD: Undecided